CLINICAL TRIAL: NCT05509660
Title: E-health Interventions for Common Mental Health Problems Among University Students in Sweden: Pilot Study of Transdiagnostic Internet-based Psychological Treatment
Brief Title: Transdiagnostic Internet Intervention to Improve Mental Health Among University Students: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Linkoeping University (Other Government); Malmö University (Other); Stockholm University (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-03599P
Record Dates: First submitted 2022-08-08; First posted 2022-08-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Psychological Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapist-guided internet-based CBT treatment with increased therapist support (Experimental): Intervention/treatment: Behavioral: 'PUMA+'
  8-week transdiagnostic CBT with therapist-support. One psychoeducation module followed by two transdiagnostic modules tailored to primary depression or anxiety symptoms, followed by three participant-choice modules, and ending with two transdiagnostic modules (acceptance; maintenance of skills learned). From mid-treatment onwards, participants will be offered increased therapist support.
  Interventions: Behavioral: PUMA+
- Therapist-guided internet-based CBT treatment with standard therapist-support (Active Comparator): Intervention/treatment: Behavioral: 'PUMA' Intervention/treatment: Behavioral: 'PUMA'
  8-week transdiagnostic CBT with therapist support. One psychoeducation module followed by two transdiagnostic modules tailored to primary depression or anxiety symptoms, followed by three participant-choice modules, and ending with two transdiagnostic modules (acceptance; maintenance of skills learned).
  Interventions: Behavioral: PUMA

INTERVENTIONS:
Behavioral: PUMA+ — Transdiagnostic CBT
  Arms: Therapist-guided internet-based CBT treatment with increased therapist support
Behavioral: PUMA — Transdiagnostic CBT
  Other Names: Transdiagnostic CBT
  Arms: Therapist-guided internet-based CBT treatment with standard therapist-support

SUMMARY:
This study comprises the pilot phase of a randomized controlled trial (NCT05085756) that will investigate the feasibility of a transdiagnostic CBT-based treatment for symptoms of depression and anxiety offered to Swedish university students. It will offer treatment to participants who have previously responded to a universal online mental health screen conducted in university setting (WHO-WMH-ICS survey).

The pilot study initially has a prospective single-group design where 30 college students with elevated depressive and/or anxiety symptoms are enrolled in 8 weeks of therapist-guided CBT treatment via the Internet. All participants included will receive treatment. Mid-treatment, participants that are judged to be at risk of treatment failure will be randomized (1:1 ratio) to either continued treatment with no change, or to receive added therapist-support intended to enhance outcome.

Pilot study outcomes include various aspects of feasibility: participant uptake, self-reported credibility and expectancy, adherence to treatment protocol and assessments, treatment satisfaction, potential adverse events, causes for premature termination of treatment, and procedures for providing additional therapist support to a subsample of participants after mid-treatment. Within-group effects for primary depression and anxiety measures will be quantified. A range of secondary measures are piloted for the subsequent randomized controlled trial. The assessment points for this study: Baseline; 8 points during treatment; post-treatment; 6-month follow-up; 12-month follow-up; 24 month follow up.

Note. This study is retrospectively registered; this registration was completed prior to any outcome data-analyses.

ELIGIBILITY:
Inclusion Criteria:

* College/university student at institution of higher education in Sweden
* Score 5-19 on the PHQ-9, and/or
* Score ≥5 on the GAD-7
* Completed baseline assessment

Exclusion Criteria:

* Pharmacotherapy for mental health issue during the past 3 weeks)
* Concurrent psychological treatment during the past 3 weeks
* Mild levels of mental ill-health (under cut-off for primary outcome measures)
* Severe levels of mental ill-health
* Suicidal ideation or plans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment Credibility and expectancy Questionnaire (CEQ). | Baseline
  Credibility/expectancy. [Feasibility and acceptability measure]
Working Alliance Inventory - Short (WAI-S) | Mid-treatment (4 weeks)
  The WAI-S is scale measuring the participants perceived working alliance with their therapist. [Feasibility and acceptability measure]
The Client Satisfaction Questionnaire-8 (CSQ-8) | Post-treatment (8 weeks)
  Treatment satisfaction [Feasibility and acceptability measure]
Treatment interest/uptake. Measured in terms of % participants who responded to the study invitation | Baseline
  Interest for intervention [Feasibility and acceptability measure]
Treatment completion/adherence. | Post-treatment (8 weeks)
  Adherence to the treatment protocol. Measured in terms of % completed modules and % of completed skills practices. [Feasibility and acceptability measure]
Assessment completion/adherence. | Post-treatment (8 weeks)
  Adherence to assessment plan (% missing data). Measured in terms of % completed measures at post-treatment. [Feasibility and acceptability measure]
Added therapist support. | Mid-treatment (4 weeks)
  Measured as % of participants who are randomized to receive additional therapist support for the remainder of the treatment period (weeks to 8).
Early treatment termination. | Post-treatment (8 weeks)
  Measured as % of participants who decide to end treatment early. This includes reporting participants' reasons for early termination, where provided. [Feasibility and acceptability measure]
Negative Effects Questionnaire (NEQ-20) | Mid-treatment (4 weeks)
  NEQ-20 investigate negative effects of psychological treatment. Total range is 0-80, with higher values representing a worse outcome. [Feasibility and acceptability measure]

SECONDARY OUTCOMES:
Patient Health Questionnaire PHQ-9 | Baseline, during treatment (weekly), post-treatment (8 weeks), follow-up at 6, 12, and 24 months
  Change in PHQ-9 at post-treatment and follow-ups as compared to baseline. Primary endpoint: Change post-treatment (8 weeks).
Generalized Anxiety Disorder scale (GAD-7) | Baseline, during treatment (weekly), post-treatment (8 weeks), follow-up at 6, 12, and 24 months
  Change in GAD-7 at post-treatment and follow-ups as compared to baseline. Primary endpoint: Change post-treatment (8 weeks).
World Health Organization Well-being questionnaire (WHO-5). | Baseline; During treatment (weekly); post-treatment (8 weeks); follow-up at 6, 12, and 24 months
  Well-being
Attitudes towards professional help (ATSPPHS) | Baseline; follow-up at 12 and 24 months
  Attitudes towards professional help
Diagnostic and Statistical Manual of Mental Disorders Cross-Cutting Symptom Measure (DSM-5 CCSM) | Baseline; mid-treatment (week 4); post-treatment (8 weeks); follow-up at 6, 12, and 24 months
  DSM-5 symptoms
Insomnia Severity Index (ISI) | Baseline; mid-treatment (4 weeks); post-treatment (8 weeks); follow-up at 6, 12, and 24 months
  Insomnia
Behavioral Activation for Depression Scale (BADS-9 | Baseline; mid-treatment (week 4); post-treatment (8 weeks); follow-up at 6, 12, and 24 months
  Behavioral Activation
Skills of Cognitive Therapy (SoCT) | Baseline; mid-treatment (4 weeks); post-treatment (8weeks); 24-month follow-up
  Cognitive Therapy skills
World Health Organization Quality of Life Scale (WHOQOL-Bref). | Baseline; follow-up at 12 and 24 months
  Quality of Life
Alcohol Use Disorders Identification Test - Consumption (AUDIT-C). | Baseline; post-treatment (8 weeks); follow-up at 6, 12, and 24 months
  Alcohol Use
Rosenberg Self-Esteem Scale (RESES) | Baseline; post-treatment (8 weeks); follow-up at 6, 12, and 24 months
  Self-Esteem
Connor-Davidson Resilience Scale. | Baseline; post-treatment (8 weeks); follow-up at 6, 12, and 24 months
  Resilience
Difficulties in Emotion-Regulation Scale (DERS-16). | Baseline; post-treatment (8 weeks); follow-up at 6, 12, and 24 months
  Emotion-Regulation
Penn-State Worry Questionnaire (PSWQ) | Baseline; post-treatment (8 weeks); follow-up at 6, 12, and 24 months
  Worry
Big Five Inventory-10 (BFI-10) | Baseline; follow-up at 12 and 24 months
  Personality
Healthcare consumption and productivity loss in patients with a psychiatric disorder (TIC-P) | Baseline; follow-up at 6, 12, and 24 months
  Healthcare consumption and productivity loss

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
Outcome data will be shared as appropriate, but primarily within the WHO-WMH-ICS consortium.

REFERENCES:
- [Background] Andersson C, Bendtsen M, Lindfors P, Molander O, Lindner P, Topooco N, Engstrom K, Berman AH. Does the management of personal integrity information lead to differing participation rates and response patterns in mental health surveys with young adults? A three-armed methodological experiment. Int J Methods Psychiatr Res. 2021 Dec;30(4):e1891. doi: 10.1002/mpr.1891. Epub 2021 Aug 21. PMID 34418224
- [Derived] Topooco N, Lindner P, Andersson C, Lindfors P, Molander O, Kraepelien M, Sundstrom C, Vlaescu G, Andersson G, Bendtsen M, Berman AH. Personalized Transdiagnostic Cognitive Behavior Therapy With Midtreatment Stepped Care to Improve Mental Health Among University Students in Sweden: Feasibility Study for a Randomized Controlled Trial. JMIR Form Res. 2026 Jan 15;10:e68698. doi: 10.2196/68698. PMID 41538789